CLINICAL TRIAL: NCT02567656
Title: A Phase I/Ib, Dose Escalation Study to Evaluate Safety and Efficacy of RP6530, a Dual PI3K δ/γ Inhibitor, in Patients With Relapsed or Refractory T-cell Lymphoma
Brief Title: Safety and Efficacy Study of a Dual PI3K Delta/Gamma Inhibitor in T-cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rhizen Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP6530-1401; 124584 (Other: Food and Drug Administration)
Record Dates: First submitted 2015-09-03; First posted 2015-10-05 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell, Cutaneous
Keywords: CTCL; PTCL; RP6530
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell, Cutaneous | interventions — tenalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): RP6530 administered orally twice a day.
  Interventions: Drug: RP6530

INTERVENTIONS:
Drug: RP6530 — Tablet starting at 200 mg
  Other Names: PI3K inhibitor

SUMMARY:
The purpose of this study is to evaluate the safety, PK and efficacy of RP6530, a dual PI3K delta/gamma inhibitor in patients with relapsed and refractory T-cell Lymphoma.

DETAILED DESCRIPTION:
Safety: Treatment-Emergent AE; Treatment-Related AE, SAE and Clinical significant AE; Dose Limiting Toxicities (DLT). PK: Peak Plasma Concentration (Cmax), Area under the plasma concentration versus time curve (AUC), Time of Maximum concentration observed (Tmax). Efficacy: Overall Response Rate (ORR), Progression Free Survival (PFS), Overall Survival (OS) and Duration of Response.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed T cell Non-Hodgkin Lymphoma (T-NHL)
* Refractory to or relapsed after at least 1 prior treatment line.
* ECOG performance status ≤2
* Patients must be ≥18 years of age
* Able to give a written informed consent.

Exclusion Criteria:

* Any cancer therapy in the last 3 weeks or limited palliative radiation <2 weeks
* Patients with HBV, HCV or HIV infection
* Previous therapy with GS-1101 (CAL-101, Idelalisib), IPI-145 (Duvelisib), TGR-1202 or any drug that specifically inhibits PI3K/ mTOR (including temsirolimus, everolimus), AKT or BTK Inhibitor (including Ibrutinib) in last 6 months
* Patients on immunosuppressive therapy including systemic corticosteroids.
* Patients with known history of liver disorders.
* Patients with uncontrolled Diabetes Type I or Type II
* Any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study.
* Women who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-09; Primary Completion 2018-03 (Actual); Study Completion 2018-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Auris Huen, MD, Principal Investigator — MD Anderson Cancer Center, Houston, Tx.
Locations (8):
- United States (8):
  - City of Hope, Duarte, California
  - Chao Family Comprehensive Cancer Center University of California Irvine, Orange, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose escalation_Cohort 1_200 mg: RP6530 administered 200 mg orally twice a day.
- Dose escalation_Cohort 2_400 mg: RP6530 administered 400 mg orally twice a day.
- Dose escalation_Cohort 3_800 mg (Fasting); Dose expansion_PTCL_800 mg (Fasting); Dose expansion_CTCL_800 mg (Fasting): RP6530 administered 800 mg orally twice a day under fasting condition
- Dose escalation_Cohort 4_800 mg (Fed): RP6530 administered 800 mg orally twice a day under fed condition
Period: Overall Study
Arm/Group | Dose escalation_Cohort 1_200 mg | Dose escalation_Cohort 2_400 mg | Dose escalation_Cohort 3_800 mg (Fasting) | Dose escalation_Cohort 4_800 mg (Fed) | Dose expansion_PTCL_800 mg (Fasting) | Dose expansion_CTCL_800 mg (Fasting)
Started | 4 | 4 | 5 | 6 | 19 | 20
Completed | 3 | 3 | 3 | 6 | 19 | 20
Not Completed | 1 | 1 | 2 | 0 | 0 | 0
Not completed — Premature discontinuation due to PD | 1 | 1 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose escalation_Cohort 1_200 mg | Dose escalation_Cohort 2_400 mg | Dose escalation_Cohort 3_800 mg (Fasting) | Dose escalation_Cohort 4_800 mg (Fed) | Dose expansion_PTCL_800 mg (Fasting) | Dose expansion_CTCL_800 mg (Fasting) | Total
Number analyzed (Participants) | 4 | 4 | 5 | 6 | 19 | 20 | 58
Age, Continuous [Median (Full Range); unit: Years] | 63.45 [47.75 to 76.58] | 65.03 [51.96 to 76.11] | 67.89 [52.11 to 70.58] | 65.86 [40.92 to 73.24] | 63.95 [53.72 to 89.55] | 67.07 [39.45 to 84.55] | 67.07 [39.45 to 89.55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 1 | 7 | 13 | 28
  Male | 1 | 2 | 3 | 5 | 12 | 7 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 4 | 4 | 8
  White | 4 | 4 | 5 | 6 | 14 | 16 | 49
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 5 | 6 | 19 | 20 | 58

OUTCOME MEASURES:

1. Primary Outcome: Safety of RP6530
Description: Number of participants with Treatment-Related Adverse Events as Assessed by CTACE v4.0
Time Frame: 28 days
Population: DLT assessment performed in patients who participated in dose escalation phase; A toxicity will be considered dose-limiting if it occurs during the first cycle (4-weeks) treatment with Tenalisib and is considered related to Tenalisib.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose escalation_Cohort 1_200 mg | Dose escalation_Cohort 2_400 mg | Dose escalation_Cohort 3_800 mg (Fasting) | Dose escalation_Cohort 4_800 mg (Fed) | Dose expansion_PTCL_800 mg (Fasting) | Dose expansion_CTCL_800 mg (Fasting)
Number analyzed (Participants) | 4 | 4 | 5 | 6 | 0 | 0
Participants
  No.of Participants with Dose Limiting Toxicities | 0 | 0 | 0 | 2 | 0 | 0
  No.of Participants without Dose Limiting Toxicitie | 4 | 4 | 5 | 4 | 0 | 0

2. Secondary Outcome: Overall Response Rate (ORR) With RP6530
Description: ORR is defined as sum of CR and PR rates, Response assessment for PTCL based on IWG criteria (Cheson 2007) and CTCL on mSWAT/Global assessment (ISCL/EORTC guideline).
Time Frame: 8 months
Population: Patients were considered for efficacy analysis as per protocol only if they had one post treatment efficacy assessment at C3D1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose escalation_Cohort 1_200 mg | Dose escalation_Cohort 2_400 mg | Dose escalation_Cohort 3_800 mg (Fasting) | Dose escalation_Cohort 4_800 mg (Fed) | Dose expansion_PTCL_800 mg (Fasting) | Dose expansion_CTCL_800 mg (Fasting)
Number analyzed (Participants) | 3 | 2 | 3 | 5 | 10 | 12
Participants | 1 | 2 | 2 | 2 | 4 | 5

3. Secondary Outcome: Duration of Response (DOR) With RP6530
Description: The time period from the response achieved in patient until the disease progression.
Time Frame: 24 months
Population: Duration of Response (DoR) is defined as the time when the measurement criteria are first met for PR or CR (whichever is reported first) until the date of documented disease progression or death. Overall number of Participants analyzed for DoR will be the participants who met response as CR or PR
Measure: Median (Full Range); unit: Days
Arm/Group | Dose escalation_Cohort 1_200 mg | Dose escalation_Cohort 2_400 mg | Dose escalation_Cohort 3_800 mg (Fasting) | Dose escalation_Cohort 4_800 mg (Fed) | Dose expansion_PTCL_800 mg (Fasting) | Dose expansion_CTCL_800 mg (Fasting)
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 4 | 5
Days | 147 [147 to 147] | 72 [29 to 115] | 313 [68 to 557] | 99 [50 to 148] | 141 [56 to 391] | 307 [67 to 588]

4. Secondary Outcome: Peak Plasma Concentration (Cmax)
Description: Peak Plasma Concentration (Cmax) of RP6530
Time Frame: Day 1 of Cycle 1
Population: Peak Plasma Concentration (Cmax) of RP6530 at Cycle 1 day 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose escalation_Cohort 1_200 mg | Dose escalation_Cohort 2_400 mg | Dose escalation_Cohort 3_800 mg (Fasting) | Dose escalation_Cohort 4_800 mg (Fed)
Number analyzed (Participants) | 4 | 4 | 5 | 6
ng/mL | 1297.65 (622.81) | 2196.65 (676.45) | 3995.68 (1392.74) | 2668.05 (1713.17)

ADVERSE EVENTS:
Time Frame: 24 months
Description: Summary of Related Treatment Emergent Adverse Events - All Patients
Arm/Group | Dose escalation_Cohort 1_200 mg | Dose escalation_Cohort 2_400 mg | Dose escalation_Cohort 3_800 mg (Fasting) | Dose escalation_Cohort 4_800 mg (Fed) | Dose expansion_PTCL_800 mg (Fasting) | Dose expansion_CTCL_800 mg (Fasting)
All-Cause Mortality (participants affected / at risk) | 0/4 | 1/4 | 1/5 | 1/6 | 3/19 | 1/20
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/5 | 0/6 | 3/19 | 3/20
Other Adverse Events (participants affected / at risk) | 4/4 | 3/4 | 5/5 | 5/6 | 11/19 | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose escalation_Cohort 1_200 mg (N=4) | Dose escalation_Cohort 2_400 mg (N=4) | Dose escalation_Cohort 3_800 mg (Fasting) (N=5) | Dose escalation_Cohort 4_800 mg (Fed) (N=6) | Dose expansion_PTCL_800 mg (Fasting) (N=19) | Dose expansion_CTCL_800 mg (Fasting) (N=20)
Pyrexia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
International normalized ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis syndrome (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose escalation_Cohort 1_200 mg (N=4) | Dose escalation_Cohort 2_400 mg (N=4) | Dose escalation_Cohort 3_800 mg (Fasting) (N=5) | Dose escalation_Cohort 4_800 mg (Fed) (N=6) | Dose expansion_PTCL_800 mg (Fasting) (N=19) | Dose expansion_CTCL_800 mg (Fasting) (N=20)
Alanine aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 2 (3) | 3 (3) | 4 (5) | 8 (13)
Aspartate aminotransferase increased (Investigations) | 1 (3) | 0 (0) | 2 (2) | 3 (10) | 4 (5) | 8 (15)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 7 (8)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 6 (6)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 5 (7)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT02567656/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT02567656/SAP_001.pdf